CLINICAL TRIAL: NCT01143818
Title: Energy, Sexual Desire and Body PropoRtions wIth AndroGel®, Testosterone 1% Gel Therapy (ESPRIT) in Hypogonadal Men
Brief Title: ESPRIT Study in Hypogonadal Men
Status: Completed | Type: Observational
Sponsor: Abbott (Industry)
Collaborators: Fovea (Other)
Responsible Party: Sponsor
Other Study IDs: S176.4.103
Record Dates: First submitted 2010-06-09; First posted 2010-06-14 (Estimated); Results first posted 2011-09-26 (Estimated); Last update posted 2011-10-17 (Estimated); Status verified 2011-10

CONDITIONS: Hypogonadism
Keywords: Male hypogonadism
MeSH Terms: conditions — Hypogonadism; Eunuchism | interventions — Testosterone

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- AndroGel (testosterone gel )1%: AndroGel is topical testosterone gel 1% (1 sachet of 5 g contains 50 mg of testosterone), 1 daily dose.
  Interventions: Drug: AndroGel (testosterone gel) 1%

INTERVENTIONS:
Drug: AndroGel (testosterone gel) 1% — AndroGel is topical testosterone gel 1% and is prescribed for once daily use.
  Other Names: Topical AndroGel; 1% AndroGel; AndroGel®

SUMMARY:
Observational study with AndroGel®, Testosterone 1% gel therapy (ESPRIT) in hypogonadal men in the community over 6 months.

DETAILED DESCRIPTION:
The objective of this study was to evaluate the efficacy and safety of AndroGel (testosterone gel) 1% following administration in community dwelling men with hypogonadism. The percent change from baseline to Month 6 in aging male symptom (AMS) assessment was the primary endpoint. Secondary endpoints were changes from baseline to Month 6 in International Index of Erectile Dysfunction (IIEF), Multidimensional Fatigue Inventory (MFI), and body mass index (BMI) assessments.

ELIGIBILITY:
Inclusion Criteria

1. Male patients >= 18 years of age
2. Hypogonadism not previously treated with testosterone
3. Testosterone deficiency confirmed clinically and biochemically
4. Being prescribed AndroGel® 1% in accordance with the local summary of product characteristics

Exclusion Criteria

1. According to the contra-indications,
2. Unwilling or unable to sign informed consent form

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community
Sampling Method: Non-Probability Sample
Enrollment: 1053 (Actual)
Dates: Start 2007-12; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Miller, PharmD, Study Director — Abbott
Locations (331):
- Canada (48):
  - Site Ref # / Investigator 59749, Burnaby, British Columbia
  - Site Ref # / Investigator 59765, Coquitlam, British Columbia
  - Site Ref # / Investigator 59742, Kamloops, British Columbia
  - Site Ref # / Investigator 59775, Kelowna, British Columbia
  - Site Ref # / Investigator 59757, Penticton, British Columbia
  - Site Ref # / Investigator 59754, Victoria, British Columbia
  - Site Ref # / Investigator 59763, Winnipeg, Manitoba
  - Site Ref # / Investigator 59762, Winnipeg, Manitoba
  - Site Ref # / Investigator 59748, Dartmouth, Nova Scotia
  - Site Ref # / Investigator 59755, Halifax, Nova Scotia
  - Site Ref # / Investigator 59753, Barrie, Ontario
  - Site Ref # / Investigator 59777, Barrie, Ontario
  - Site Ref # / Investigator 59744, Burlington, Ontario
  - Site Ref # / Investigator 59766, Corunna, Ontario
  - Site Ref # / Investigator 59773, Greater Sudbury, Ontario
  - Site Ref # / Investigator 59751, Greater Sudbury, Ontario
  - Site Ref # / Investigator 59752, Hamilton, Ontario
  - Site Ref # / Investigator 59764, Jarvis, Ontario
  - Site Ref # / Investigator 59774, Lindsay, Ontario
  - Site Ref # / Investigator 59768, London, Ontario
  - Site Ref # / Investigator 59776, Markham, Ontario
  - Site Ref # / Investigator 59759, Mississauga, Ontario
  - Site Ref # / Investigator 59761, Mississauga, Ontario
  - Site Ref # / Investigator 54484, North York, Ontario
  - Site Ref # / Investigator 59760, Ottawa, Ontario
  - Site Ref # / Investigator 59747, Pickering, Ontario
  - Site Ref # / Investigator 59750, Sarnia, Ontario
  - Site Ref # / Investigator 59745, Scarborough Village, Ontario
  - Site Ref # / Investigator 59771, Sherbrooke, Ontario
  - Site Ref # / Investigator 59772, Stoney Creek, Ontario
  - Site Ref # / Investigator 59756, Toronto, Ontario
  - Site Ref # / Investigator 59758, Toronto, Ontario
  - Site Ref # / Investigator 59767, Welland, Ontario
  - Site Ref # / Investigator 59743, Windsor, Ontario
  - Site Ref # / Investigator 59788, Beauceville, Quebec
  - Site Ref # / Investigator 59780, Grand-Mère, Quebec
  - Site Ref # / Investigator 59785, L'lle Perrot, Quebec
  - Site Ref # / Investigator 59769, Montreal, Quebec
  - Site Ref # / Investigator 59746, Mount Royal, Quebec
  - Site Ref # / Investigator 59781, Québec, Quebec
  - Site Ref # / Investigator 59770, Saint-Ambroise, Quebec
  - Site Ref # / Investigator 59779, Saint-Ambroise, Quebec
  - Site Ref # / Investigator 59787, Saint-Hyacinthe, Quebec
  - Site Ref # / Investigator 59782, Saint-Lambert-de-Lauzon, Quebec
  - Site Ref # / Investigator 59786, Saint-Nicolas, Quebec
  - Site Ref # / Investigator 59784, Ste-Marthe-sur-le-Lac, Quebec
  - Site Ref # / Investigator 59783, Trois-Rivières, Quebec
  - Site Ref # / Investigator 59778, Ville Mont-Royal, Quebec
- Croatia (28):
  - Site Ref # / Investigator 59628, Dubrovnik
  - Site Ref # / Investigator 59627, Karlovac
  - Site Ref # / Investigator 59540, Osijek
  - Site Ref # / Investigator 59626, Pula
  - Site Ref # / Investigator 59554, Rijeka
  - Site Ref # / Investigator 59622, Rijeka
  - Site Ref # / Investigator 59623, Rijeka
  - Site Ref # / Investigator 59624, Rijeka
  - Site Ref # / Investigator 59629, Rijeka
  - Site Ref # / Investigator 59550, Split
  - Site Ref # / Investigator 59551, Split
  - Site Ref # / Investigator 59552, Split
  - Site Ref # / Investigator 59553, Split
  - Site Ref # / Investigator 59625, Split
  - Site Ref # / Investigator 59536, Zagreb
  - Site Ref # / Investigator 59537, Zagreb
  - Site Ref # / Investigator 59538, Zagreb
  - Site Ref # / Investigator 59539, Zagreb
  - Site Ref # / Investigator 59541, Zagreb
  - Site Ref # / Investigator 59542, Zagreb
  - Site Ref # / Investigator 59543, Zagreb
  - Site Ref # / Investigator 59544, Zagreb
  - Site Ref # / Investigator 59545, Zagreb
  - Site Ref # / Investigator 59546, Zagreb
  - Site Ref # / Investigator 59547, Zagreb
  - Site Ref # / Investigator 59548, Zagreb
  - Site Ref # / Investigator 59549, Zagreb
  - Site Ref # / Investigator 54485, Zagreb
- Germany (32):
  - Site Ref # / Investigator 59864, Bad Kreuznach
  - Site Ref # / Investigator 59867, Bad Schönborn
  - Site Ref # / Investigator 59889, Berlin
  - Site Ref # / Investigator 59884, Cologne
  - Site Ref # / Investigator 59879, Duisburg
  - Site Ref # / Investigator 59868, Erkrath
  - Site Ref # / Investigator 59862, Erlangen
  - Site Ref # / Investigator 59872, Essen
  - Site Ref # / Investigator 59886, Essen
  - Site Ref # / Investigator 59888, Frankfurt
  - Site Ref # / Investigator 59881, Freiburg im Breisgau
  - Site Ref # / Investigator 59861, Garmisch-Patenkirchen
  - Site Ref # / Investigator 59882, Gelsenkirchen
  - Site Ref # / Investigator 59876, Giessen
  - Site Ref # / Investigator 59883, Halle
  - Site Ref # / Investigator 59880, Hamburg
  - Site Ref # / Investigator 59870, Kamp-Lintfort
  - Site Ref # / Investigator 59860, Landstuhl
  - Site Ref # / Investigator 59877, Marburg
  - Site Ref # / Investigator 59866, München
  - Site Ref # / Investigator 59863, Münster
  - Site Ref # / Investigator 59874, Neuss
  - Site Ref # / Investigator 59890, Nieder-Olm
  - Site Ref # / Investigator 59873, Nienburg
  - Site Ref # / Investigator 59887, Osnabrück
  - Site Ref # / Investigator 59878, Paderborn
  - Site Ref # / Investigator 59875, Plön
  - Site Ref # / Investigator 59871, Saarlouis
  - Site Ref # / Investigator 59885, Schwelm
  - Site Ref # / Investigator 59869, Seligenstadt
  - Site Ref # / Investigator 54486, Warendorf
  - Site Ref # / Investigator 59865, Weiden
- Kuwait (6):
  - Site Ref # / Investigator 59631, Ad Dasmah
  - Site Ref # / Investigator 54487, Ahmandi
  - Site Ref # / Investigator 59633, Al Ahmadi
  - Site Ref # / Investigator 59634, As Sālimīyah
  - Site Ref # / Investigator 59630, Bayān
  - Site Ref # / Investigator 59632, Bayān
- Romania (29):
  - Site Ref # / Investigator 59488, Arad
  - Site Ref # / Investigator 59483, Brasov
  - Site Ref # / Investigator 59461, Bucharest
  - Site Ref # / Investigator 59460, Bucharest
  - Site Ref # / Investigator 59455, Bucharest
  - Site Ref # / Investigator 59459, Bucharest
  - Site Ref # / Investigator 59454, Bucharest
  - Site Ref # / Investigator 54489, Bucharest
  - Site Ref # / Investigator 59456, Bucharest
  - Site Ref # / Investigator 59458, Bucharest
  - Site Ref # / Investigator 59457, Bucharest
  - Site Ref # / Investigator 59462, Bucharest
  - Site Ref # / Investigator 59465, Cluj-Napoca
  - Site Ref # / Investigator 59473, Cluj-Napoca
  - Site Ref # / Investigator 59464, Cluj-Napoca
  - Site Ref # / Investigator 59463, Cluj-Napoca
  - Site Ref # / Investigator 59466, Cluj-Napoca
  - Site Ref # / Investigator 59475, Cluj-Napoca
  - Site Ref # / Investigator 59479, Iași
  - Site Ref # / Investigator 59476, Iași
  - Site Ref # / Investigator 59477, Iași
  - Site Ref # / Investigator 59478, Iași
  - Site Ref # / Investigator 59480, Iași
  - Site Ref # / Investigator 59484, Sibiu
  - Site Ref # / Investigator 59482, Târgu Mureş
  - Site Ref # / Investigator 59481, Târgu Mureş
  - Site Ref # / Investigator 59485, Timișoara
  - Site Ref # / Investigator 59487, Timișoara
  - Site Ref # / Investigator 59486, Timișoara
- Russia (75):
  - Site Ref # / Investigator 59891, Kazan'
  - Site Ref # / Investigator 59695, Kazan'
  - Site Ref # / Investigator 59643, Kemerovo
  - Site Ref # / Investigator 59697, Kemerovo
  - Site Ref # / Investigator 59893, Khabarovsk
  - Site Ref # / Investigator 59654, Khabarovsk
  - Site Ref # / Investigator 59897, Krasnodar
  - Site Ref # / Investigator 59900, Krasnodar
  - Site Ref # / Investigator 59675, Krasnoyarsk
  - Site Ref # / Investigator 59903, Krasnoyarsk
  - Site Ref # / Investigator 59678, Moscow
  - Site Ref # / Investigator 59651, Moscow
  - Site Ref # / Investigator 59902, Moscow
  - Site Ref # / Investigator 59688, Moscow
  - Site Ref # / Investigator 59698, Moscow
  - Site Ref # / Investigator 59665, Moscow
  - Site Ref # / Investigator 59896, Moscow
  - Site Ref # / Investigator 59689, Moscow
  - Site Ref # / Investigator 59650, Moscow
  - Site Ref # / Investigator 59648, Moscow
  - Site Ref # / Investigator 59646, Moscow
  - Site Ref # / Investigator 59649, Moscow
  - Site Ref # / Investigator 59662, Moscow
  - Site Ref # / Investigator 59645, Naberezhnye Chelny
  - Site Ref # / Investigator 59638, Nizhny Novgorod
  - Site Ref # / Investigator 59677, Nizhny Novgorod
  - Site Ref # / Investigator 59668, Nizhny Novgorod
  - Site Ref # / Investigator 59693, Novosibirsk
  - Site Ref # / Investigator 59656, Novosibirsk
  - Site Ref # / Investigator 59895, Novosibirsk
  - Site Ref # / Investigator 59694, Novosibirsk
  - Site Ref # / Investigator 59641, Penza
  - Site Ref # / Investigator 59637, Penza
  - Site Ref # / Investigator 59657, Penza
  - Site Ref # / Investigator 59636, Rostov-on-Don
  - Site Ref # / Investigator 59699, Rostov-on-Don
  - Site Ref # / Investigator 59655, Rostov-on-Don
  - Site Ref # / Investigator 59667, Rostov-on-Don
  - Site Ref # / Investigator 54490, Saint Petersburg
  - Site Ref # / Investigator 59691, Saint Petersburg
  - Site Ref # / Investigator 59640, Saint Petersburg
  - Site Ref # / Investigator 59676, Saint Petersburg
  - Site Ref # / Investigator 59642, Saint Petersburg
  - Site Ref # / Investigator 59700, Saint Petersburg
  - Site Ref # / Investigator 59679, Saint Petersburg
  - Site Ref # / Investigator 59658, Saint Petersburg
  - Site Ref # / Investigator 59672, Samara
  - Site Ref # / Investigator 59661, Saratov
  - Site Ref # / Investigator 59666, Saratov
  - Site Ref # / Investigator 59663, Tolyatti
  - Site Ref # / Investigator 59905, Tolyatti
  - Site Ref # / Investigator 59653, Tolyatti
  - Site Ref # / Investigator 59692, Tomsk
  - Site Ref # / Investigator 59690, Tomsk
  - Site Ref # / Investigator 59673, Tomsk
  - Site Ref # / Investigator 59669, Ufa
  - Site Ref # / Investigator 59670, Ufa
  - Site Ref # / Investigator 59659, Ufa
  - Site Ref # / Investigator 59652, Ufa
  - Site Ref # / Investigator 59660, Vladivostok
  - Site Ref # / Investigator 59901, Vladivostok
  - Site Ref # / Investigator 59639, Vladivostok
  - Site Ref # / Investigator 59635, Volgograd
  - Site Ref # / Investigator 59892, Volgograd
  - Site Ref # / Investigator 59696, Voronezh
  - Site Ref # / Investigator 59906, Voronezh
  - Site Ref # / Investigator 59671, Voronezh
  - Site Ref # / Investigator 59894, Voronezh
  - Site Ref # / Investigator 59664, Yaroslavl
  - Site Ref # / Investigator 59899, Yaroslavl
  - Site Ref # / Investigator 59674, Yaroslavl
  - Site Ref # / Investigator 59647, Yekaterinburg
  - Site Ref # / Investigator 59904, Yekaterinburg
  - Site Ref # / Investigator 59898, Yekaterinburg
  - Site Ref # / Investigator 59644, Yekaterinburg
- Saudi Arabia (64):
  - Site Ref # / Investigator 59398, Abhā
  - Site Ref # / Investigator 59405, Dammam
  - Site Ref # / Investigator 59406, Dammam
  - Site Ref # / Investigator 59388, Dammam
  - Site Ref # / Investigator 59446, Dammam
  - Site Ref # / Investigator 59424, Hofouf
  - Site Ref # / Investigator 59429, Hofouf
  - Site Ref # / Investigator 59395, Jeddah
  - Site Ref # / Investigator 59423, Jeddah
  - Site Ref # / Investigator 59404, Jeddah
  - Site Ref # / Investigator 59809, Jeddah
  - Site Ref # / Investigator 59396, Jeddah
  - Site Ref # / Investigator 59437, Jeddah
  - Site Ref # / Investigator 59441, Jeddah
  - Site Ref # / Investigator 59444, Jeddah
  - Site Ref # / Investigator 59385, Jeddah
  - Site Ref # / Investigator 59435, Jeddah
  - Site Ref # / Investigator 59807, Jeddah
  - Site Ref # / Investigator 59806, Jeddah
  - Site Ref # / Investigator 59390, Jeddah
  - Site Ref # / Investigator 59443, Jeddah
  - Site Ref # / Investigator 59397, Jeddah
  - Site Ref # / Investigator 59392, Jeddah
  - Site Ref # / Investigator 59805, Jubail
  - Site Ref # / Investigator 54491, Khamis Mushait
  - Site Ref # / Investigator 59402, Khamis Mushait
  - Site Ref # / Investigator 59804, Khamis Mushait
  - Site Ref # / Investigator 59387, Khobar
  - Site Ref # / Investigator 59426, Khobar
  - Site Ref # / Investigator 59438, Khobar
  - Site Ref # / Investigator 59453, Khobar
  - Site Ref # / Investigator 59383, Madinah
  - Site Ref # / Investigator 59384, Madinah
  - Site Ref # / Investigator 59428, Madinah
  - Site Ref # / Investigator 59439, Madinah
  - Site Ref # / Investigator 59808, Madinah
  - Site Ref # / Investigator 59386, Mecca
  - Site Ref # / Investigator 59393, Mecca
  - Site Ref # / Investigator 59403, Mecca
  - Site Ref # / Investigator 59448, Riyadh
  - Site Ref # / Investigator 59389, Riyadh
  - Site Ref # / Investigator 59432, Riyadh
  - Site Ref # / Investigator 59440, Riyadh
  - Site Ref # / Investigator 59400, Riyadh
  - Site Ref # / Investigator 59399, Riyadh
  - Site Ref # / Investigator 59422, Riyadh
  - Site Ref # / Investigator 59451, Riyadh
  - Site Ref # / Investigator 59425, Riyadh
  - Site Ref # / Investigator 59427, Riyadh
  - Site Ref # / Investigator 59430, Riyadh
  - Site Ref # / Investigator 59452, Riyadh
  - Site Ref # / Investigator 59449, Riyadh
  - Site Ref # / Investigator 59433, Riyadh
  - Site Ref # / Investigator 59442, Riyadh
  - Site Ref # / Investigator 59447, Riyadh
  - Site Ref # / Investigator 59401, Riyadh
  - Site Ref # / Investigator 59394, Riyadh
  - Site Ref # / Investigator 59436, Riyadh
  - Site Ref # / Investigator 59391, Tabuk
  - Site Ref # / Investigator 59407, Tabuk
  - Site Ref # / Investigator 59434, Tabuk
  - Site Ref # / Investigator 59445, Tabuk
  - Site Ref # / Investigator 59450, Tabuk
  - Site Ref # / Investigator 59431, Yanbu
- Slovenia (16):
  - Site Ref # / Investigator 59800, Celje
  - Site Ref # / Investigator 59802, Celje
  - Site Ref # / Investigator 59798, Celje
  - Site Ref # / Investigator 54492, Ljubljana
  - Site Ref # / Investigator 59791, Ljubljana
  - Site Ref # / Investigator 59792, Ljubljana
  - Site Ref # / Investigator 59793, Ljubljana
  - Site Ref # / Investigator 59794, Ljubljana
  - Site Ref # / Investigator 59797, Ljubljana
  - Site Ref # / Investigator 59799, Ljubljana
  - Site Ref # / Investigator 59789, Maribor
  - Site Ref # / Investigator 59790, Maribor
  - Site Ref # / Investigator 59795, Maribor
  - Site Ref # / Investigator 59796, Maribor
  - Site Ref # / Investigator 59801, Maribor
  - Site Ref # / Investigator 59803, Novo Mesto
- United Arab Emirates (33):
  - Site Ref # / Investigator 59502, Abu Dhabi
  - Site Ref # / Investigator 59506, Abu Dhabi
  - Site Ref # / Investigator 59513, Abu Dhabi
  - Site Ref # / Investigator 59524, Abu Dhabi
  - Site Ref # / Investigator 59526, Abu Dhabi
  - Site Ref # / Investigator 59528, Abu Dhabi
  - Site Ref # / Investigator 59516, Ajman
  - Site Ref # / Investigator 59519, Ajman
  - Site Ref # / Investigator 59514, Alain
  - Site Ref # / Investigator 59532, Alain
  - Site Ref # / Investigator 59534, Dubai
  - Site Ref # / Investigator 59523, Dubai
  - Site Ref # / Investigator 59508, Dubai
  - Site Ref # / Investigator 54493, Dubai
  - Site Ref # / Investigator 59504, Dubai
  - Site Ref # / Investigator 59505, Dubai
  - Site Ref # / Investigator 59509, Dubai
  - Site Ref # / Investigator 59511, Dubai
  - Site Ref # / Investigator 59517, Dubai
  - Site Ref # / Investigator 59518, Dubai
  - Site Ref # / Investigator 59521, Dubai
  - Site Ref # / Investigator 59525, Dubai
  - Site Ref # / Investigator 59529, Dubai
  - Site Ref # / Investigator 59531, Dubai
  - Site Ref # / Investigator 59533, Dubai
  - Site Ref # / Investigator 59510, Ras al-Khaimah
  - Site Ref # / Investigator 59515, Ras al-Khaimah
  - Site Ref # / Investigator 59522, Sharjah city
  - Site Ref # / Investigator 59530, Sharjah city
  - Site Ref # / Investigator 59507, Sharjah city
  - Site Ref # / Investigator 59512, Sharjah city
  - Site Ref # / Investigator 59535, Sharjah city
  - Site Ref # / Investigator 59527, Sharjah city

REFERENCES:
- See also: Related Info — http://dailymed.nlm.nih.gov/dailymed/drugInfo.cfm?id=23151&CFID

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants enrolled in this study were newly-diagnosed for hypogonadism and treatment naive to testosterone preparations. A total of 1053 participants were enrolled but only 1049 were treated with AndroGel.
Pre-assignment Details: AndroGel (testosterone gel) 1% was prescribed according to the regional Summary of Product Characteristics with a starting dose of 50 mg testosterone/day (packaged as 1 sachet of 50 mg). Testosterone was applied once daily.
Groups:
- AndroGel (Testosterone Gel) 1%: Topical testosterone gel 1% (1 sachet of 5 g contains 50 mg of testosterone), 1 daily dose. All participants who received at least 1 dose of study drug are included in the safety analysis set.
Period: Overall Study
Arm/Group | AndroGel (Testosterone Gel) 1%
Started | 1049 (A total of 1053 participants were enrolled but only 1049 received study drug.)
Completed | 799
Not Completed | 250

BASELINE CHARACTERISTICS:
Arm/Group | AndroGel (Testosterone Gel) 1%
Number analyzed (Participants) | 1049
Age Continuous [Mean (Standard Deviation); unit: years] | 53 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1049
Region of Enrollment [Number; unit: Participants]
  Canada | 338
  Russian Federation | 267
  Croatia | 134
  Germany | 91
  Slovenia | 87
  Saudi Arabia | 68
  Romania | 54
  United Arab Emirates | 10

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline to Month 6 in Aging Male Symptoms (AMS) in Mean Total Score
Description: The Aging Male Symptoms (AMS) test is self-administered and designed to assess symptoms of aging with a rating from none (0) to extremely severe (5) for 17 items from psychological (5 items), somatic (7 items), and sexual (5 items) categories. Total scores range from 17 (minimum) to 85 (maximum). The AMS total score was reported at baseline and at Month 6 and represented the sum of all the items. The percent change from baseline was calculated as the [(AMS value at Month 6 - AMS value at baseline)/baseline value] x 100.
Time Frame: Baseline to Month 6
Population: The full analysis set included all participants in the safety analysis set who had an Aging Male Symptoms (AMS) score available at baseline and Month 6.
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | AndroGel (Testosterone Gel) 1%
Number analyzed (Participants) | 712
Percent Change | -29.0 (22.6)

2. Secondary Outcome: Percent Change From Baseline to Month 6 in the International Index of Erectile Function (IIEF) Total Score
Description: The International Index of Erectile Function (IIEF) test is a validated 15 question assessment designed to measure changes in erectile function (6 items), orgasmic function (2 items), sexual desire (2 items), intercourse satisfaction (3 items), and overall satisfaction (2 items). The scores ranged from 0 to 5 on each item with a lower score indicating greater dysfunction. A total IIEF score of 0 (minimum) to 75 (maximum) was possible and represented the sum of all the items at baseline and Month 6. The percent change = [(IIEF value at Month 6-IIEF baseline value)/IIEF baseline value]x 100.
Time Frame: Baseline to Month 6
Population: The full analysis set included all participants in the safety analysis set who had an IIEF score available at baseline and Month 6.
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | AndroGel (Testosterone Gel) 1%
Number analyzed (Participants) | 651
Percent Change | 115.7 (226.3)

3. Secondary Outcome: Percent Change From Baseline to Month 6 in the Multidimensional Fatigue Inventory (MFI) Total Score
Description: The MFI is a 20-item self-reported instrument designed to measure fatigue. Five scales measure different modes of fatigue: general fatigue (4 items), physical fatigue (4 items), mental fatigue (4 items), reduced motivation (4 items), and reduced activity items (4 items). The scores for each item range from 1 to 5. Each subscale includes 4 items with 5-point Likert scales and subscale scores range from 4 to 20 with a higher score indicating greater fatigue. The percent change=[(MFI value at Month 6-MFI value at baseline)/MFI baseline value] X 100.
Time Frame: Baseline to Month 6
Population: The full analysis set included all participants in the safety analysis set who had an MFI score available at baseline and Month 6.
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | AndroGel (Testosterone Gel) 1%
Number analyzed (Participants) | 655
Percent Change | -21.5 (33.5)

4. Secondary Outcome: Percent Change From Baseline to Month 6 in Body Mass Index (BMI)
Description: The BMI was measured in kg/m^2 and was reported at baseline and at the Month 6. BMI = weight (kg)/[(height (m) x height (m)] and was measured to 1 decimal point precision.
Time Frame: Baseline to Month 6
Population: The full analysis set included all participants in the safety analysis set who had BMI available at baseline and Month 6.
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | AndroGel (Testosterone Gel) 1%
Number analyzed (Participants) | 611
Percent Change | -2.38 (5.75)

ADVERSE EVENTS:
Time Frame: All reported adverse events are treatment-emergent and are defined as events that started or worsened at or after the first administration of AndroGel and ended before or at treatment completion. Only suspected adverse drug reactions were collected.
Description: Treatment-emergent adverse events that were not serious occurred in 64 patients. None of the adverse events occured at a frequency threshold of >=5%. Therefore, no adverse events were reported.
Arm/Group | AndroGel (Testosterone Gel) 1%
Serious Adverse Events (participants affected / at risk) | 3/1049
Other Adverse Events (participants affected / at risk) | 0/1049
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AndroGel (Testosterone Gel) 1% (N=1049)
Angina pectoris (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Hypertension (Vascular disorders) | 1
Nausea (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Abbott requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. Abbott requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Abbott needs to secure patent or proprietary protection.